CLINICAL TRIAL: NCT00245180
Title: Primordial Prevention of Overweight in American Indian Children
Brief Title: Preventing American Indian Children From Becoming Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 239; U01HL081624 (NIH)
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2006-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- control (No Intervention): Primary and secondary data collected as in intervention arm. Dental screenings will be done once a year as a service.
  Interventions: Behavioral: Diet; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Diet
Behavioral: Exercise

SUMMARY:
The purpose of this study is to establish an intervention to keep American Indian/Alaskan Native (AI/AN) children from becoming overweight.

DETAILED DESCRIPTION:
BACKGROUND:

AI/AN children have overweight rates that are 18 to 30 percent higher than the general American population of children. Adult obesity has early antecedents, and data show that eating and physical activity behaviors are formed and set as early as 3 years of age, through primary socialization within families. Yet there are few, if any, obesity prevention programs that target children younger than 3 years of age.

DESIGN NARRATIVE:

This is a community-partnered randomized study to prevent early childhood overweight in AI/AN children. A birth cohort of about 780 children from six Indian communities born over a period 18 months will be randomized by community to either a control (3 communities) or intervention condition (3 communities). The intervention comprises a community-wide intervention coupled with individualized family counseling to improve nutrition and physical activity in infants and toddlers. Nutrition goals are to increase breastfeeding initiation and sustainability, limit sugared beverages for infants and toddlers, and make healthful choices during weaning and solid food introduction. Physical activity goals include promoting motor development, limiting video/TV viewing, and creating play opportunities for infants and toddlers. Intervention approaches and methods used in the pilot study on which this project is based will be combined with new formative data collected at the beginning of the project to enhance the intervention's feeding and physical activity components. Each component in the community-wide interventions will be collaboratively designed with the tribes, and tailored to each community's needs. Trained peer counselors will deliver the family interventions, during a series of 12 cluster visits, each covering a different developmental stage of the infant/toddler.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had uncomplicated pregnancies
* Women who agree to have their child enrolled in the study and followed for 30 months
* Women who are not planning to leave their area within 2 years of study start

Exclusion Criteria:

* Women whose children have a serious illness known to affect normal growth

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 577 (Actual)
Dates: Start 2006-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
BMI | birth, 6,12,18, and 24 months

SECONDARY OUTCOMES:
feeding | 0-24 months
  Breastfeeding, (initiation and maintenance), introduction of solids.

CONTACTS AND LOCATIONS:
Overall Officials: Njeri Karanja, Principal Investigator — Kaiser Foundation Hospitals